CLINICAL TRIAL: NCT03707821
Title: Design Validation of Senofilcon A With New UV-blocking Additive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6305
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- senofilcon A TEST Lens (Experimental): Subjects between 18 to 49 years of age that are habitual wearers of spherical soft contact lenses will be randomized into the TEST Lens for the duration of the clinical study.
  Interventions: Device: senofilcon A TEST Lens
- senofilcon A CONTROL Lens (Active Comparator): Subjects between 18 to 49 years of age that are habitual wearers of spherical soft contact lenses will be randomized into the CONTROL Lens for the duration of the clinical study.
  Interventions: Device: senofilcon A CONTROL Lens

INTERVENTIONS:
Device: senofilcon A TEST Lens — JJVC Investigational Contact Lens
  Arms: senofilcon A TEST Lens
Device: senofilcon A CONTROL Lens — Acuvue Oasys
  Arms: senofilcon A CONTROL Lens

SUMMARY:
This is a 2-visit, multi-site, partially subject-masked, 2-arm parallel, controlled, randomized and dispensing trial. Subjects will be randomized to one of two study lenses for the entire duration of the study. The study lenses will be worn for a period of 2 weeks each in a bilateral fashion.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Between 18 and 49 (inclusive) years of age at the time of informed consent.
  4. Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them when needed for near vision.
  5. The subject is a current spherical soft contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week wear time over the last 30 days by self-report.
  6. Subjects must be able and willing to wear the study lenses at least 6 hours a day, a minimum of 5 days per week.
  7. Subjects must own a wearable pair of distance spectacles.
  8. The subject's vertex-corrected spherical equivalent distance refraction must be in the range of -1.00 to -6.00 D (inclusive) in each eye.
  9. The subject's refractive cylinder must be 0.00 to -1.00 D (inclusive) in each eye.
  10. The subject must have a spherocylindrical best corrected distance Snellen visual acuity of 20/25+3 or better in each eye.

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
  2. Any active or ongoing systemic disease (e.g., Sjögren's Syndrome), infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis).
  3. Subjects taking suspect oral medications for less than one year.
  4. Any prescribed or over the counter (OTC) ocular medication.
  5. Any known hypersensitivity or allergic reaction to Optifree® PureMoist® multi-purpose care solution or Eye-Cept® rewetting drop solution.
  6. Toric, extended wear, monovision or multi-focal contact lens correction.
  7. Any previous or planned (during the course of the study) ocular surgery (e.g., PRK, LASIK, etc.).
  8. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
  9. Participation in clinical trials involving the Test lens within 3 months prior to study enrollment.
  10. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  11. Binocular vision abnormality or strabismus by self-report or prior medical history.
  12. History of recurrent corneal erosions, herpetic keratitis, or pathological dry eye.
  13. Any active ocular allergies, infections or other ocular abnormalities (entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma) that the investigator determines may interfere with the outcomes of this study or otherwise contraindicate participation in the study.
  14. Any Grade 2 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA Slit Lamp Classification Scale.
  15. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar) within the past 3 years of otherwise successful contact lens wear.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 253 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - James T. Fujimoto, OD, Cupertino, California
  - Maitland Vision Center, Maitland, Florida
  - Tallahassee Eye Center, Tallahassee, Florida
  - Eyecare Associates LLP, Bloomington, Illinois
  - Kannarr Eye Care, Pittsburg, Kansas
  - ProCare Vision Centers, Granville, Ohio
  - Professional Vision Care, Inc, Westerville, Ohio
  - Bradley Hines, OD, Memphis, Tennessee
  - Frazier Vision, Inc, Tyler, Texas
  - Ziegler Leffingwell Eyecare, New Berlin, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 253 subjects were enrolled into this study. Of those 2 subjects failed to meet all eligibility criteria and 251 subjects were dispensed a study lens. of the dispensed subjects 248 completed the study while 3 subjects were discontinued.
Groups:
- Test: Subjects that wore the Test lens in both eyes during the entire duraiton of the study.
- Control: Subjects that wore the Control lens in both eyes throughout the entire duration of the study.
Period: Overall Study
Arm/Group | Test | Control
Started | 125 | 126
Completed | 123 | 125
Not Completed | 2 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Unsatisfactory Visual Response | 1 | 0
Not completed — Unsatisfactory Lens Fitting | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: All subjects dispensed the Control lens in both eyes throughout the entire duration of the study.
- Total: Total of all reporting groups
Arm/Group | Test | Control | Total
Number analyzed (Participants) | 125 | 126 | 251
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.5 (6.59) | 31.7 (6.73) | 31.1 (6.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 84 | 169
  Male | 40 | 42 | 82
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 10 | 11 | 21
  Black or African American | 0 | 4 | 4
  White | 115 | 109 | 224
  Other | 0 | 2 | 2
Region of Enrollment [Number; unit: Participants]
  United States | 125 | 126 | 251

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort Score
Description: Overall comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patientexperience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 2-Week Follow-up Evlauation
Population: All subjects that completed the study without a major protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Control: Subjects that wore the Control lens in both eyes during the entire duraiton of the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 122 | 124
Units on a Scale | 64.7 (21.33) | 62.6 (23.38)
Statistical Analysis 1: Comparison: Test vs Control; It was calculated that 224 participants randomized in a 1:1 fashion between the two lens types would have at least 80% power to detect a 5 points difference in mean overall comfort at he 2-week follow-up. Sample size was determined using Stroup's Method (alpha=0.05); Test type: Non-Inferiority — A non-inferiority margin of -5 points was used. This margin is based on a 10% shift in the distribution of CLUE scores. Non-inferiority was declared in the lower limit of the 95% credible interval was above 5; Bayesian normal random-effects; A 95% Credible Interval for the Posterior mean difference between the Test and Control was used to test for non-inferiority; Mean Difference (Net) = 3.3, 95% CI 2-sided [-2.0 to 8.5], Standard Deviation 2.65 — Mean difference was calculated as Test minus Control

2. Primary Outcome: Vision Satisfaction in Bright Lighting
Description: Vision satisfaction in bright light was assessed using the individual item" I was satisfied with the quality of my vision in bright lighting" from the CLUE™ questionnaire. This item used the response scale, 1: Strongly Disagree, 2: Disagree, 3: Neither Agree nor Disagree, 4: Agree and 5: Strongly Agree. CLUE is the Contact Lens User Experience™ questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The Proportion of responses in each category were reported for each lens type.
Time Frame: 2-Week Follow-up Evaluation
Population: Subjects that completed all study visits without a major protocol deviation impacting a primary endpoint.
Measure: Number; unit: Percentage of subjects
Arm/Group | Test | Control
Number analyzed (Participants) | 122 | 124
Percentage of subjects
  Strongly Agree | 30.3 | 19.4
  Agree | 59.0 | 58.1
  Neither Agree nor Disagree | 6.6 | 12.9
  Disagree | 4.1 | 8.1
  Strongly Disagree | 0 | 0.8
Statistical Analysis 1: Comparison: Test vs Control; It was calculated that 40 participants randomized in a 1:1 fashion between the two lens types would have at least 80% power to detect a 10% difference in proportion of subjects that reported at higher rating (Strongly Agree and Agree) with the Test compared to the Control lens at the 2-week follow-up. Sample size was determined using simulation-based methods (alpha=0.05); Test type: Non-Inferiority — A cumulative odds ratio non-inferiority margin of 2 was used. This margin is based on a 10% difference if the proportion of subjects that report a higher rating/experience; Bayesian random -effects model; A 95% Credible Interval for the Posterior proportion mean difference between the Test and Control was used to test for non-inferiority; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [0.02 to 0.15], Standard Deviation 0.034 — mean difference was calculated as Test minus Control

3. Primary Outcome: Distance Visual Acuity
Description: Distance visual acuity was assessed by eye using LogMAR visual acuity at 4 meters using an ETDRS chart under high illumination high contrast conditions (room illumination > 400 lux and chart luminance 120-200 cd/m2) at the 2-week follow-up for each subject eye. Lower values of logMAR indicate better vision, where a score of 0.0 equates to 20/20 snellen vision. The average visual acuity for each lens was reported.
Time Frame: 2-Week Follow-up Evlauation
Population: Subjects that completed all study visits without a major protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Test | Control
Number analyzed (Participants) | 122 | 124
Number analyzed (eyes) | 244 | 248
logMAR | -0.131 (0.0913) | -0.107 (0.0861)
Statistical Analysis 1: Comparison: Test vs Control; It was calculated that 30 participants randomized in a 1:1 fashion between the two lens types would have at least 80% power to detect a 0.05 difference in LogMAR visual acuity at the 2-week follow-up. Sample size was determined using simulations methods for repeated measures; Test type: Non-Inferiority — A non-inferiority margin of 0.05 points was used. This margin corresponds to a half line difference; Bayesian Normal Random effects model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.04 to -0.01], Standard Deviation 0.008 — Mean difference was calculated as Test minus Control

4. Primary Outcome: Contact Lens Fitting Acceptance Rate
Description: Acceptable lens fit will be assessed at all study visits (scheduled and unscheduled) for each subject eye. Fit acceptance rate will be based on the lens fit acceptance of eyes wearing the Test lens only. Fit acceptance is a binary response where Y=1 if lens fit is acceptable and Y=0 otherwise. Unacceptable is defined as unacceptable if any one of the following criteria:
  * limbal exposure at primary gaze or with extreme eye movement;
  * edge lift;
  * excessive movement in primary up gaze;
  * insufficient movement in all three of the following conditions: primary gaze, up gaze, and push up test.
  Eyes with multiple unacceptable fitting events will be counted only once. Fit rates of the Control lens will also be collected but are not a primary endpoint.
Time Frame: Up to 2-Week Follow-up
Population: All subjects that were dispsensed a study lens.
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Test | Control
Number analyzed (Participants) | 125 | 126
Number analyzed (eyes) | 250 | 252
Percentage of eyes | 99.2 | 100
Statistical Analysis 1: Comparison: Test; It was calculated that 100 participants were required to show that the acceptable lens fitting for the Test lens would be superior to 90% with at least 80% power. Sample size was determined using simulations methods for repeated measures; Test type: Superiority — A superiority margin of 90% was used. Lower limit of 95% credible interval was compared to 90%; Bayesian Beta-Binomial Model; model for correlated data; Mean Percentage of Acceptable Fitting = 99.5, 95% CI 2-sided [98.5 to 100], Standard Deviation 0.38

5. Primary Outcome: Number of Grade 3 or Higher Slit Lamp Findings
Description: Slit Lamp Findings (SLF) were assessed using a biomicroscope and was graded using the FDA grading scale (Grade: 0, 1,2, 3 and 4) with grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e. Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). Slit Lamp Findings will be assessed for each subject eye at all study visits (schedule and unscheduled). SLF is a binary response where Y=1 for at least one Grade 3 or 4 slit lamp finding. The percentage of eyes with Grade 3 or higher slit lamp findings will be analyzed and will include corneal infiltrates. Eyes with multiple events will be counted only once. The number of eyes with SLF with grade 3 or higher by lens was reported.
Time Frame: Up to 2-Week Follow-up Evlauation
Population: All subjects that were dispensed a study lens.
Measure: Number; unit: Number of eyes
Units Other Than Participants: eyes
Arm/Group | Test | Control
Number analyzed (Participants) | 125 | 126
Number analyzed (eyes) | 250 | 252
Number of eyes | 0 | 0
Statistical Analysis 1: Comparison: Test vs Control; It was calculated that 224 participants randomized in a 1:1 fashion between the two lens types would have at least 80% power to detect 5% difference between the Test and Control lens with respect to the proportion of eyes with Grade 3 or higher slit lamp findings across all study visits. Sample size was determined using simulations methods. Sample size for this study was primarily driven by the slit lamp findings; Test type: Non-Inferiority — A non-inferiority margin of 5% was used. Upper limit of the 95% credible interval was compared to 5%; Bayesian beta-binomial model; model for correlated data; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.007 to 0.008], Standard Deviation 0.0036 — mean difference was calculated as Test minus Control

6. Secondary Outcome: Overall Handling Score
Description: Overall handling was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patientexperience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 2-Week Follow-up Evlauation
Population: All subjects that completed the study without a major protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Test | Control
Number analyzed (Participants) | 122 | 124
Units on a Scale | 70.9 (17.24) | 68.7 (18.55)
Statistical Analysis 1: Comparison: Test vs Control; Sample Size was based on primary endpoints only; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Bayesian normal random-effects; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 2.5, 95% CI 2-sided [-1.3 to 6.3], Standard Deviation 1.94 — Mean difference was calculated as Test minus Control

7. Secondary Outcome: Overall Quality of Vision Score
Description: Overall quality of vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patientexperience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 2-Week Follow-up Evlauation
Population: All subjects that completed the study without a major protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Test | Control
Number analyzed (Participants) | 122 | 124
Units on a Scale | 66.4 (19.19) | 60.9 (22.33)
Statistical Analysis 1: Comparison: Test vs Control; Sample Size was based on primary endpoints only; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Bayesian normal random-effects; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 8.03, 95% CI 2-sided [3.48 to 12.54], Standard Deviation 2.295 — Mean difference was calculated as Test minus Control

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 2-Weeks per subject.
Groups:
- Control: Subjects that wore the Control lens at any point during the study.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/126
Other Adverse Events (participants affected / at risk) | 0/125 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT03707821/SAP_000.pdf
  • Study Protocol (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT03707821/Prot_001.pdf